CLINICAL TRIAL: NCT05037006
Title: A Comparison of Three Different Doses of Neostigmine on the Reversal of Cisatracurium-induced Moderate Neuromuscular Blockade in Patients Under Sevoflurane or TIVA Anesthesia.
Brief Title: Three Different Doses of Neostigmine on the Reversal of Cisatracurium-induced Moderate Neuromuscular Blockade
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 50358321.5.0000.5373
Record Dates: First submitted 2021-08-12; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Neuromuscular Blockade; Neuromuscular Blockade, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of randomized computer-generated numbers (www.random.org) will be used for this purpose. No surgeon, members of the nursing team, anesthesiologist involved in anesthesia or data collection will be aware of the dose of neostigmine to be administered. The type of anesthesia (inhalation or venous) will not be covered. An anesthesiologist not involved in the study will be responsible for preparing the solution containing neostigmine and atropine (diluted with saline solution until complete 20 mL) according to the group to which each patient belongs. Syringes (20 mL) will be similar and identified only with a label with the word "reversal".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group I-30 (Experimental): Inhalational anesthesia and reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
  Interventions: Drug: Sevoflurane - Neostigmine 30
- Group I-50 (Experimental): Inhalational anesthesia and reversal with neostigmine 50 mcg/kg and atropine 25 mcg/kg
  Interventions: Drug: Sevoflurane - Neostigmine 50
- Group I-70 (Experimental): Inhalational anesthesia and reversal with neostigmine 70 mcg/kg and atropine 35 mcg/kg
  Interventions: Drug: Sevoflurane - Neostigmine 70
- Group V-30 (Experimental): Intravenous anesthesia and reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
  Interventions: Drug: TIVA - Neostigmine 30
- Group V-50 (Experimental): Intravenous anesthesia and reversal with neostigmine 50 mcg/kg and atropine 25 mcg/kg
  Interventions: Drug: TIVA - Neostigmine 50
- Group V-70 (Experimental): Intravenous anesthesia and reversal with neostigmine 70 mcg/kg and atropine 35 mcg/kg
  Interventions: Drug: TIVA - Neostigmine 70

INTERVENTIONS:
Drug: Sevoflurane - Neostigmine 30 — Neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOFc 3
  Other Names: Inhalational anesthesia
  Arms: Group I-30
Drug: Sevoflurane - Neostigmine 50 — Neostigmine 50 mcg/kg and atropine 25 mcg/kg when TOFc 3
  Other Names: Inhalational anesthesia
  Arms: Group I-50
Drug: Sevoflurane - Neostigmine 70 — Neostigmine 70 mcg/kg and atropine 35 mcg/kg when TOFc 3
  Other Names: Inhalational anesthesia
  Arms: Group I-70
Drug: TIVA - Neostigmine 30 — Neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOFc 3
  Other Names: TIVA
  Arms: Group V-30
Drug: TIVA - Neostigmine 50 — Neostigmine 50 mcg/kg and atropine 25 mcg/kg when TOFc 3
  Other Names: TIVA
  Arms: Group V-50
Drug: TIVA - Neostigmine 70 — Neostigmine 70 mcg/kg and atropine 35 mcg/kg when TOFc 3
  Other Names: TIVA
  Arms: Group V-70

SUMMARY:
The aim of the present study will be to evaluate by means of a prospective randomized clinical trial, the time required for the reversal of moderate neuromuscular blockade (NMB) (Train-of-four count = 3; TOFc 3) to Train-of-four ratio (TOFr) > 0.9 and TOFr = 1.0 after administration of different doses of neostigmine (30, 50 and 70 mcg/kg) in patients undergoing general anesthesia with propofol or sevoflurane. In addition, the probability of NMB reversal in less than 10 minutes or 15 minutes after neostigmine administration will be registered.

DETAILED DESCRIPTION:
METHODS

After the approval of the Research Ethics Committee of the Faculty of Medical and Health Sciences of Pontificia University Catholic of Sao Paulo (PUC-SP), patients submitted to nose or ear surgeries at Santa Lucinda Hospital and able to participate in this clinical, prospective, and randomized trial will be evaluated. The following will be included: patients aged between 18 and 65 years old, physical status according to the American Society of Anesthesiologists I and II, submitted to general anesthesia. Exclusion criteria will be: (i) refusal to participate in the study; (ii) presence of kidney, liver or neuromuscular disease; (iii) contraindication to the use of any of the drugs used in the study or (iv) body mass index (BMI) ≥ 30. Patients will be randomly distributed into one of 6 groups according to the type of anesthesia (inhalational or venous) and the dose of neostigmine used to reverse NMB:

* Group I-30: inhalational anesthesia and reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
* Group I-50: inhalational anesthesia and reversal with neostigmine 50 mcg/kg and atropine 25 mcg/kg
* Group I-70: inhalational anesthesia and reversal with neostigmine 70 mcg/kg and atropine 35 mcg/kg
* Group V-30: intravenous anesthesia and reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
* Group V-60: intravenous anesthesia and reversal with neostigmine 50 mcg/kg and atropine 25 mcg/kg
* Group V-70: intravenous anesthesia and reversal with neostigmine 70 mcg/kg and atropine 35 mcg/kg.

For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of randomized computer-generated numbers (www.random.org) will be used for this purpose. No surgeon, members of the nursing team, anesthesiologist involved in anesthesia or data collection will be aware of the dose of neostigmine to be administered. The type of anesthesia (inhalation or venous) will not be covered. An anesthesiologist not involved in the study will be responsible for preparing the solution containing neostigmine and atropine (diluted with saline solution until complete 20 mL) according to the group to which each patient belongs. Syringes (20 mL) will be similar and identified only with a label with the word "reversal".

STUDY SEQUENCE

Anesthesia

After entry into the operating room, all patients will be monitored with cardioscopy, noninvasive blood pressure, pulse oximetry and, after tracheal intubation, with capnography. Venous access will be obtained on one of the upper limbs. After pre-oxygenation, anesthetic induction and maintenance will be as follows:

1. Group I-30, I-50 and I-70 - Induction with remifentanil at a dose of 0.5 mcg/kg/min for 3 minutes, followed by a maintenance dose of 0.3 mcg/kg/min. Propofol bolus (2.0 mg/kg) followed by maintenance with sevoflurane 2% diluted in O2/air flow (60%) 2L/min.
2. Group V-30, V-50 and V-70 - Induction with remifentanil at a dose of 0.5 mcg/kg/min for 3 minutes, followed by maintenance dose of 0.3 mcg/kg/min. Bolus propofol (2.0 mg/kg) followed by infusion at the rate of 4 to 6 mg/kg/h.

For both groups, cisatracúrio (0.1 mg/kg) will be administered before tracheal intubation, which will be performed when T1 was less than 5%. Ventilation will be controlled, with tidal volume and respiratory rate adjusted for the maintenance of PETCO2 between 30 and 40 mmHg. When there is a suspect of inadequate anesthesia plan, the infusion rate of propofol or sevoflurane will be increased and if adequacy is not sufficient, the infusion rate of remifentanil will be increased. Patients who have a decrease in systolic blood pressure (SBP) greater than 30% or heart rate (HR) less than 50 bpm will be treated with ephedrine (10 mg) and atropine (0.5 mg), respectively. Hydration will be performed with 0.9% saline solution (500 ml in the first 30 minutes and 2 mL/kg/min the following hours). The central temperature will be maintained above 35oC and peripheral (tenar eminence of the monitored palm) above 32o C. Reversal of NMB will be performed when TOFc 3 by administration of the previously prepared solution.

Monitoring of neuromuscular blockade NMB will be monitored by acceleromyography method (TOF Watch SX®;¬ Schering-Plough) as recommended for use in clinical research. 9 The acceleration transducer will be fixed on the volar side of the distal phalanx of the thumb. Venous access and blood pressure cuff will be positioned on the opposite arm to the limb used for NMB monitoring. After cleaning the skin in the path of the ulnar nerve in the forearm, the electrodes will be positioned at the height of the wrist with a distance between 3 to 6 cm between them. Calibration will be performed after automatically after a 50 Hz tetanus stimulus for 5 seconds. The stimulation (Train-of-Four-TOF) will be applied every 15 seconds for 2 minutes before cisatracúrio is given. No additional doses of NMB will be administered. Once the third response to the TOF is obtained, a dose of neostigmine (30, 50 or 70 mcg/kg) will be administered and the time for until the TOF reaches values equal to 0.9 and 1.0 will be recorded. The primary outcome will be the time required for the reversal of moderate NMB (TOF=3) up to TOF = 0.9 and TOF = 1.0. In addition, the probability of reversion of NMB will be evaluated in less than 10 minutes or 15 minutes after the administration of different doses of neostigmine in patients undergoing intravenous or inhalational anesthesia. The sample size will be based on a previous study that determined the need for 12 patients per group to detect with a power of 90% and alpha error of 5% a difference between groups equal to or greater than 1.3 standard deviations. 10 Considering possible losses, 90 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients physical status according to the American Society of Anesthesiologists I and II
* submitted to nose or ear surgeries under general anesthesia

Exclusion Criteria:

* Refusal to participate in the study
* Presence of kidney, liver or neuromuscular disease
* Contraindication to the use of any of the drugs used in the study
* Body mass index (BMI) ≥ 30.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Reversal from TOFc 3 to TOFr 1.0 | Time from neostigmine administration up to 60 minutes
  Time required the appearance of the third response to TOF stimulation to complete NMB reversal
Reversal from TOFc 3 to TOFr 0.9 | Time from neostigmine administration up to 60 minutes
  Time required the appearance of the third response to TOF stimulation to TOFr 0.9

SECONDARY OUTCOMES:
Probability of complete NMB reversal in less than 10 minutes | Time from neostigmine administration up to 60 minutes
  The probability of NMB reversal in less than 10 minutes after neostigmine administration will be evaluated
Probability of complete NMB reversal in less than 15 minutes | Time from neostigmine administration up to 60 minutes
  The probability of NMB reversal in less than 15 minutes after neostigmine administration will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, MD, Principal Investigator — Pontificia Catholic University of São Paulo
Locations (1):
- Santa Lucina Hospital, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No